CLINICAL TRIAL: NCT04778514
Title: A Randomized, Crossover Study Comparing Adherence, Preference + Acceptability of a Dual Prevention Pill (DPP) Capsule Containing PrEP + an Oral Contraceptive Versus Two Separate Pills in Women at Risk of HIV in Harare, Zimbabwe
Brief Title: A Crossover Acceptability Study Assessing a DPP Capsule for HIV and Pregnancy Prevention
Acronym: 952
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Population Council (Other)
Collaborators: University of Zimbabwe (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: Protocol #952
Record Dates: First submitted 2021-02-25; First posted 2021-03-03 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: HIV Infections; Contraception
MeSH Terms: conditions — HIV Infections | interventions — Contraceptives, Oral, Combined; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Intervention Model Description: A randomized, open-label, parallel group, 2-way crossover study A total of 24 weeks (6 28-day menstrual cycles); 3 cycles of DPP capsule (12 weeks); 3 cycles of 2 separate tablets (PrEP and COC tablets; 12 weeks)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sequence 1 (Other): This arm is a single, over-encapsulated DPP containing PrEP (200 mg of emtricitabine [FTC], 300 mg of tenofovir disoproxil fumarate [TDF]) and a COC (30 mcg of ethinyl estradiol [EE], 150 mcg of levonorgestrel [LNG]) taken once daily for three 28-day cycles followed by PrEP (FTC/TDF) and a COC (EE/LNG) taken daily for three 28-day cycles.
  Interventions: Drug: Dual Prevention Pill; Drug: PrEP and combined oral contraceptive (COC) as two separate tablets
- Sequence 2 (Other): This arm is two separate tablets (PrEP [FTC/TDF] and COC [EE/LNG]) taken once daily for three 28-day cycles followed by single, over-encapsulated DPP containing PrEP (FTC/TDF) and a COC (EE/LNG) taken once daily for three 28-day cycles.
  Interventions: Drug: Dual Prevention Pill; Drug: PrEP and combined oral contraceptive (COC) as two separate tablets

INTERVENTIONS:
Drug: Dual Prevention Pill — a single over-encapsulated DPP containing a PrEP tablet and a COC
  Other Names: DPP
Drug: PrEP and combined oral contraceptive (COC) as two separate tablets — PrEP tablet and a COC as two separate tablets
  Other Names: Truvada; Zinnia F

SUMMARY:
The study design is a single-site, two-arm, randomized, open-label crossover trial in 30 AGYW aged 16-24 in Chitungwiza (Harare), Zimbabwe. The aim of the study is to assess the acceptability of, preference for, and adherence to a single DPP capsule containing one PrEP tablet and one COC tablet compared to two separate tablets (FTC/TDF and EE/LNG), each taken for three consecutive menstrual cycles for a total of 24 weeks among current COC users.

DETAILED DESCRIPTION:
We will conduct a randomized, open-label, parallel group, 2-way crossover study among approximately 30 girls and young women (AGYW) aged 16-24 years old to compare adherence, preference, acceptability and safety of a single dual prevention pill (DPP) containing Truvada and the generic COC, Zinnia F (Regimen A), versus Truvada and Zinnia F taken separately (Regimen B). All participants must already be using COCs for at least 3 months prior to screening and must plan to continue using them for at least one year. We are enrolling women who are already using COCs because we believe they are most likely to be interested in a daily oral MPT. Furthermore, we would like participants who are already accustomed to COCs so that they can have a clearer sense of how PrEP - whether taken separately or in the DPP - makes them feel.

Prior to the commencement of the study, the Population Council procured and qualified all study drugs required for the crossover study, including: bulk pills (Truvada and Zinnia F) for encapsulation, COC pill packs, and bottles of Truvada. Under the guidance of the Council's clinical and regulatory groups, PCI Pharma (Rockford, IL, USA) over-encapsulated Truvada and Zinnia F according to Good Manufacturing Practices. The over-encapsulated pills were then blister packaged, pouched, and kitted for distribution to participants.

The DPP regimen (A) consists of a kit containing 4 pouches with a 28-day supply of over-encapsulated pills; 21 pink and white capsules will contain Truvada over-encapsulated together with a COC; the other 7 capsules, corresponding to the 7 placebo days in a COC pill pack, will be white and will contain Truvada only. The provider counseling manual will emphasize the fact that unlike a COC pill pack where 7 pills are placebo, all of the pills in the regimen contain Truvada, so it will be important to take them for all 28 days. For Regimen B, participants will receive a 28-day blister pack of Zinnia F, as is currently marketed, with 21 active pills and 7 placebo pills. Truvada will be dispensed in bottles of 30 pills, as is currently marketed. Participants will be instructed to take one Truvada tablet and one COC table daily for 28 days.

After providing written informed consent (or assent, with parental consent, for non-emancipated 16-17-year-old girls), women will be screened for eligibility. Participants can be enrolled if they are sexually-active (defined as having had penile-vaginal sex with a male ≤3 months before screening), currently using a COC that was started ≥3 months before screening, HIV-negative (based on HIV rapid test at screening), not-pregnant (based on hCG urine test at screening), have no contraindications for PrEP or COCs, and are in good health based on medical history and vital signs. PrEP screening will follow the standard of care in Zimbabwe, which recommends testing for Hepatitis B, hepatitis C, complete blood count (CBC), blood creatinine levels, pregnancy, and STIs. Women who test positive for pregnancy or HIV will be referred per the local standard of care. Participants who test positive for a curable STI will be treated and enrolled. Participants who are eligible will be scheduled for an enrollment visit on Day 0 of their menstrual cycle.

At enrollment, women will be randomly assigned to one of two sequences of the two regimens, with all women using both regimens by the end of the crossover study. The Population Council study biostatistician created the randomization scheme using Statistical Analysis Software (SAS/STAT) version 9.4 (SAS Institute Inc., Cary, North Carolina) with a 1:1 allocation using permutated block sizes. 15 participants will be assigned to Sequence 1: DPP capsules (Regimen A) in period 1, and two separate tablets (Regimen B) in period 2, and 15 participants will be assigned to Sequence 2: Regimen B in period 1 and Regimen A in period 2. Randomization will be in blocks of 10, with 5 participants assigned to each sequence in each of the 3 blocks. Participants will use each regimen for 3 28-day menstrual cycles and will then switch to the second regimen at their crossover visit.

Participants will attend a total of up to 8 clinic visits including Screening, Enrollment and monthly follow up visits for up to 7 months. No wash-out period is required between regimens. At Visit 1, prior to initiating product use, participants will be asked to complete a baseline behavioral interview and will be asked which regimen they think they will prefer. At all other visits, participants will complete behavioral interviews (approximately 30 minutes) about adherence and acceptability. All behavioral interviews will be conducted using computer assisted self-interviewing (CASI), which has been shown to elicit more truthful reporting than face-to-face interviewing. At the end of the Crossover period, participants will complete their final CASI interview, in which they will be asked to 1) state their preference for the DPP or 2 separate pills; 2) to qualify the strength of their preference on a scale of 1-10; All of the participants who complete the study and anyone who withdraws early will be asked to take part in an in-depth interview to explore qualitatively reasons for continuation and discontinuation, as well as the influence of partners, family, support structures, side effects, provider interactions and other factors on cMPT choice and adherence.

At all follow up visits, women will be tested for HIV and pregnancy, report adverse events (AEs) and have a clinical exam, if necessary, and respond to a structured questionnaire via computer assisted self-interview (CASI) with questions about acceptability, preference, and adherence. At the end of the Crossover period, women will be asked to state which regimen they prefer. Accrual is estimated to take approximately 6 months from first participant enrolling to last participant completing the study. We will assess and compare PrEP acceptability and adherence by regimen and overall, and we will investigate if specific socio-ecological factors (e.g., individual-, partner-, family-, and clinic-level) are associated with adherence and acceptability. We will also explore facilitators and barriers to use by conducting in-depth interviews with a subset of willing participants who complete the study and any women who withdraws early. Furthermore, because we assume people are predisposed to judge a specific regimen or technology based on initial impressions, we will assess if pre-use preferences are associated with actual experiences and preferences after using each regimen.

At each visit, women will be tested for pregnancy and HIV and will provide a blood sample for DBS to assess drug levels/adherence to PrEP. Adverse events will be recorded during the study, although no pharmacokinetic interactions are expected because there are no drug-drug interactions between the reverse transcriptase inhibitors tenofovir and emtricitabine, and the contraceptive hormones levonorgestrel and ethinyl estradiol. In addition, the side effects profiles of the two products are similar; the most commonly reported side-effects for both Truvada® and COCs are headache and nausea. Since we are recruiting women who are already using COCs, participants will already be accustomed to side-effects of COCs. Participants will be encouraged to contact or visit the clinic with questions or concerns between visits.

Rapid HIV testing will be done at screening, in accordance with local guidelines. Pregnancy will be tested based on hCG levels in urine. DBS collected from enrolled participants will be sent to the University of Cape Town where tenofovir disoproxil fumarate (TDF) drug levels will be measured to evaluate adherence based on expected levels for daily use.

Quantitative and qualitative behavioral collection instruments will adhere to our theoretical framework for assessing acceptability, with questions adapted from previous HIV-prevention studies, as relevant. In-depth interview guides will be developed from instruments used in previous PrEP introduction studies and tailored for this study.

Quantitative data from the CASI behavioral interviews will be saved at the site in .csv (comma separated value) format and shared with Population Council weekly via encrypted zip files. Clinical data collected from participants, including background demographics; medical and pregnancy history; vital signs; concomitant medications; AEs; enrollment and termination dates; and records of returned unused pills will be entered into REDCap, an electronic data system. Data from CASI interviews, eCRFs and DBS analysis will be formatted into SAS data sets for analysis. Descriptive statistics (frequencies, mean, standard deviation, range) will be used to summarize data collected and to characterize differences in participants assigned to each Sequence. Modeling will be used to assess the impact of background characteristics on adherence, preference and acceptability.

PC conducted site initiation and training for the crossover study in collaboration with UZ-CTRC, which has extensive experience implementing qualitative and quantitative HIV prevention research studies. The Population Council and site coordinator have weekly teleconferences and the full teams are meeting monthly during data collection to discuss and resolve any issues as they occur. The PC clinical research associate will make periodic monitoring trips during data collection to ensure the safety of participants and adherence to the protocol. The PC team will also review data collected on a weekly basis.

ELIGIBILITY:
Inclusion Criteria:

1. Age 16 through 24 years old (inclusive) at Screening, verified per site-specific SOPs.
2. Able and willing to provide informed consent per site SOPs. (If under the legal age of consent [18 years old] be able to provide informed assent and obtain parental or guardian consent, to be screened for and to enroll in the study.)
3. Fluent in spoken Shona and/or English.
4. Able and willing to provide adequate locator information, as defined in site SOPs.
5. Able and willing to comply with all study procedures, including being comfortable taking the study products as evident by nurse/clinician-observed swallowing at Screening of a large Vitamin capsule that is of similar size to the study products.
6. Post-menarche, per participant report at Screening.
7. Sexually active, defined as having had penile-vaginal sex with a male within the 3 months before Screening (per self-report).
8. At moderate to high risk of HIV infection based on clinician assessment.
9. Considers herself to be at moderate to high risk of HIV acquisition based on self-assessment.
10. Currently using COCs for contraception and has been using them for at least 3 months prior to Screening.
11. HIV-negative per rapid test at Screening and Enrolment per site-specific SOP.
12. Negative pregnancy test at Screening and Enrolment.
13. Negative for chlamydia, gonorrhea, trichomoniasis, and syphilis at Screening; women who test positive at Screening may be treated and enrolled.
14. Hepatitis B surface antigen and Hepatitis C negative per blood test at Screening.
15. Normal estimated creatinine clearance (eCrCl) ≥ 60 ml/min per blood test at Screening.

Exclusion Criteria:

1. Currently using emtricitabine (FTC) or tenofovir (TDF) at Screening (per self-report)
2. Intends to become pregnant within the next 12 months.
3. Intolerance, adverse reaction, or laboratory abnormality associated with PrEP use in the past.
4. Use of PEP within 3 months of Screening (per self-report).
5. Breastfeeding < 6 months postpartum (per self-report).
6. Less than 6 weeks (≤42 days) postpartum and not breastfeeding (per self-report).
7. History of deep vein thrombosis / pulmonary embolism (self-report) or history of thrombophlebitis or thromboembolic disorders at Screening (per self-report or medical records).
8. Prolonged immobilization (self-report).
9. Known thrombogenic mutation/complicated valvular disease (per self-report).
10. History of cerebro-vascular or coronary artery disease reported at Screening.
11. Ischemic heart disease (per self-report).
12. Systemic lupus erythematosus with positive or unknown antiphospholipid antibodies (per self-report).
13. Migraines with aura
14. History of undiagnosed abnormal genital bleeding reported at Screening.
15. Current breast cancer or within 5 years of past breast cancer (per self-report) or history of carcinoma of the breast or other estrogen-dependent neoplasia reported at Screening.
16. Diabetes with nephropathy, retinopathy, or neuropathy (per self-report).
17. Diabetes for > 20 years (per self-report).
18. Symptomatic gall bladder disease (per self-report).
19. Severe cirrhosis (per self-report).
20. Liver tumor (per self-report).
21. Any other condition the clinician feels would jeopardize the health and wellbeing of the participant.

Ages: 16 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2022-12-07 (Actual); Primary Completion 2023-09-11 (Actual); Study Completion 2023-09-11 (Actual)

PRIMARY OUTCOMES:
To determine preference for taking a single DPP capsule versus 2 separate tablets (PrEP and COC) once daily among women after using each regimen for three 28-day cycles. | at study completion (approximately 24 weeks)
  Proportion of women who prefer the DPP (Regimen A) vs 2 separate tablets (Regimen B) after using each regimen for 3 28-day cycles, per self-report on computer-assisted self-interviewing (CASI).
To assess the acceptability of taking the DPP capsule versus two separate tablets once daily to prevent HIV and unintended pregnancy among women who use each regimen for three 28-day cycles. | At the 3 and 6 month visits.
  Acceptability scores by regimen and overall, per a quantitative acceptability questionnaire via CASI.

SECONDARY OUTCOMES:
To assess and compare daily adherence to PrEP for six 28-day cycles among AGYW when taken in the DPP capsule (Regimen A) or as a separate tablet (Regimen B) via a biomarker. | Monthly, through 24 weeks
  TFV-DP drug levels in dried blood spots (DBS).
To assess and compare self-reported adherence to PrEP for six 28-day cycles among AGYW when taken in the DPP capsule (Regimen A) or as a separate tablet (Regimen B). | Monthly, through 24 weeks
  Proportion of PrEP doses taken compared to total number of doses expected per self-report based on a CASI questionnaire.
To assess and compare adherence to the DPP (Regimen A) vs PrEP as a separate tablet (Regimen B) each used for 3 28-day cycles by pill count. | Monthly, through 24 weeks
  Proportion of DPP and PrEP doses taken compared to total number of doses expected per pill count.
To explore if socio-ecological factors, product characteristics and product use experiences are associated with adherence to PrEP whether taken as part of the DPP capsule or as a separate tablet. | Baseline and monthly through 24 weeks
  Results of multivariate modeling indicating which, if any, factors are associated with adherence.
To explore if socio-ecological factors, product characteristics and product use experiences are associated with acceptability of the DPP and of 2 separate tablets. | at study completion (approximately 24 weeks)
  Results of multivariate modeling indicating which, if any, factors are associated with acceptability.
To qualitatively understand barriers and facilitators to product use and adherence. | at study completion (approximately 24 weeks)
  Results of thematic qualitative data analysis from in-depth interviews with participants at study exit focusing on facilitators and barriers of product use and adherence.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Friedland, MPH, Study Director — Population Council
Locations (1):
- University of Zimbabwe Clinical Trials Research Centre (UZ-CTRC), Belgravia, Harare, Zimbabwe

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mgodi NM, Burnett-Zieman JB, Murombedzi C, Dandadzi A, Gatsi V, Musara P, Matimbira S, Mavemwa G, Jambaya J, Chidemo T, Plagianos M, Haddad LB, Bruce IV, Mathur S, Friedland BA. A Dual Prevention Pill for HIV & Pregnancy Prevention: A Pilot Study Among Adolescent Girls and Young Women in Zimbabwe. AIDS Behav. 2025 Nov 18. doi: 10.1007/s10461-025-04909-2. Online ahead of print. PMID 41251867
- [Derived] Friedland BA, Mgodi NM, Palanee-Phillips T, Mathur S, Plagianos MG, Bruce IV, Lansiaux M, Murombedzi C, Musara P, Dandadzi A, Reddy K, Ndlovu N, Zulu SK, Shale LR, Zieman B, Haddad LB. Assessing the acceptability of, adherence to and preference for a dual prevention pill (DPP) for HIV and pregnancy prevention compared to oral pre-exposure prophylaxis (PrEP) and oral contraception taken separately: protocols for two randomised, controlled, cross-over studies in South Africa and Zimbabwe. BMJ Open. 2024 Mar 12;14(3):e075381. doi: 10.1136/bmjopen-2023-075381. PMID 38479746